CLINICAL TRIAL: NCT03715101
Title: A Clinical Study to Evaluate Pharmacokinetic, Pharmacodynamic, and Pharmacogenomic Characteristics of Rosuvastatin in the Elderly After Multiple Administration of Rosuvastatin
Brief Title: A Clinical Study to Evaluate PK, PD, and PG of Rosuvastatin in the Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, MD, PhD, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rosuvastatin_Elderly
Record Dates: First submitted 2017-07-19; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Elderly
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rosuvastatin 20 mg PO (Experimental): Rosuvastatin 20 mg daily for 21 days
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Open-label, one-sequence, multiple administration
  Other Names: Rosuvastatin 20 mg

SUMMARY:
A clinical study to evaluate pharmacokinetic, pharmacodynamic, and pharmacogenomic characteristics of Rosuvastatin in the elderly after multiple administration of Rosuvastatin

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects aged 65 - 85 years
* A body mass index (BMI) in the range of 18.5 kg/m2 - 27.0 kg/m2.
* Good health based on complete medical history, physical examinations, vital signs, electrocardiography (ECG), and clinical laboratory evaluations.

Exclusion Criteria:

* Subjects who have clinically significant disease of cardiovascular, respiratory, renal, endocrinological, hematological, gastrointestinal, neurological(central nervous system), psychiatric disorders or malignant tumor
* Subject judged not eligible for study participation by investigator

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters (Tmax; time to reach maximum plasma concentration) of rosuvastatin | Day 21 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour, 12 hour, 24 hour
  Pharmacokinetic evaluation
Pharmacokinetic parameters (Cmax; peak plasma concentration) of rosuvastatin | Day 21 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour, 12 hour, 24 hour
  Pharmacokinetic evaluation
Pharmacokinetic parameters (AUC; area under the concentration-time curve) of rosuvastatin | Day 21 0 hour, 1 hour, 2 hour, 3 hour, 4 hour, 5 hour, 8 hour, 12 hour, 24 hour
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
lipid panel (low-density lipoprotein cholesterol in mg/dL) | Day 1 0 hour, Day 11 0 hour, Day 22 0 hour
  Pharmacodynamic evaluation
lipid panel (high-density lipoprotein cholesterol in mg/dL) | Day 1 0 hour, Day 11 0 hour, Day 22 0 hour
  Pharmacodynamic evaluation
lipid panel (Triglyceride in mg/dL) | Day 1 0 hour, Day 11 0 hour, Day 22 0 hour
  Pharmacodynamic evaluation
lipid panel (Total cholesterol in units of mg/dL) | Day 1 0 hour, Day 11 0 hour, Day 22 0 hour
  Pharmacodynamic evaluation
lipid metabolites | Day -1 0 hour, Day 21 0 hour
  Metabolites evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, Principal Investigator — South Korea Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: Undecided